CLINICAL TRIAL: NCT07046780
Title: A Multicenter, Prospective, Non-Interventional Real-World Study of Iparomlimab and Tuvonralimab Injection (QL1706) in the Treatment of Locally Advanced or Metastatic Solid Tumors
Status: Not yet recruiting | Type: Observational
Sponsor: PENG YUAN (Other)
Responsible Party: Sponsor-Investigator, PENG YUAN, Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Other Study IDs: NCC5416
Record Dates: First submitted 2025-06-23; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Solid Tumor Cancer; Metastatic Solid Tumors; Locally Advanced

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation group: Patients treated with Iparomilimab and Tuvonralimab in the real world
  Interventions: Drug: Observation arm

INTERVENTIONS:
Drug: Observation arm — To observe the efficacy and safety of Iparomilimab and Tuvonralimab in the treatment of patients with solid tumors in the real world

SUMMARY:
This study is a prospective, observational, real-world, multi-center study planning to enroll 90 patients. The study will observe and document patients' actual clinical practices in receiving Iparomlimab and Tuvonralimab Injection (QL1706). The primary objectives are to evaluate the safety and effectiveness of Iparomlimab and Tuvonralimab Injection (QL1706) in treating locally advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* 1) Histologically or cytologically confirmed locally advanced or metastatic solid tumors with disease progression (radiographic or clinical) after ≥1 line of prior standard therapy, unsuitable for/intolerant to standard therapy. Includes but not limited to: Gastrointestinal tumors (colorectal cancer, hepatocellular carcinoma, esophageal cancer, biliary tract cancer, pancreatic cancer, gastric cancer), Breast cancer, Non-small cell lung cancer (NSCLC), Small cell lung cancer (SCLC), Soft tissue sarcoma;
* 2) ECOG performance status 0-2;
* 3) ≥1 measurable lesion per RECIST v1.1 ;
* 4) Adequate organ function meeting ALL criteria below:

  1. Hematology (without transfusion/G-CSF support within 7 days):

     Absolute neutrophil count (ANC) ≥1.5×10⁹/L Platelets ≥100×10⁹/L Hemoglobin ≥90 g/L
  2. Biochemistry :

     Total bilirubin (TBIL) ≤2×ULN ALT/AST ≤2.5×ULN (≤5×ULN if liver metastases present) Serum creatinine (Cr) ≤1.5×ULN Albumin ≥28 g/L
  3. Urinalysis :

     Urine protein <2+ (dipstick) If protein ≥2+, 24h urinary protein ≤1.0 g
  4. Coagulation (without anticoagulants):

PT/APTT/INR ≤1.5×ULN

* 5) Life expectancy ≥12 weeks;
* 6) Contraception : Females of childbearing potential or males with partners of childbearing potential must use effective contraception during treatment and for 6 months post-treatment;
* 7) Signed informed consent and protocol compliance.

Exclusion Criteria:

* 1) Tumor-Related Conditions

  1. Known CNS metastases (except those radiologically stable ≥4 weeks after radiotherapy);
  2. Other malignancies within past 5 years, excluding:

     Cured basal/squamous cell skin cancer Localized low-risk prostate cancer Cervical/breast carcinoma in situ
  3. Severe bone lesions from metastatic disease, including:

     Uncontrolled bone pain Pathologic fractures at critical sites (within 6 months) or impending spinal cord compression;
  4. Uncontrolled effusions requiring recurrent drainage (pleural/pericardial/ascites), per investigator assessment.
* 2) Prior Anti-tumor Therapy

  1. Prior systemic therapy with CTLA-4 inhibitors or other ICIs;
  2. Any anti-tumor treatment within 4 weeks before first dose, including:

     Surgery/chemotherapy/palliative radiotherapy to non-target lesions/hormonal/targeted/biologic/immunotherapy;
  3. Treatment-related toxicities not recovered to CTCAE grade ≤1 (exceptions: alopecia/platinum-induced neuropathy ≤ grade 2).
* 3) Comorbidities & History

  1. Arterial thromboembolism within 6 months (MI/unstable angina/stroke/TIA);
  2. Symptomatic heart failure (NYHA class III-IV), unstable angina, or uncontrolled arrhythmia;
  3. Severe pulmonary disease : ILD/COPD/symptomatic bronchospasm;
  4. Active uncontrolled infection (≥CTCAE grade 2), including:

     HIV Active HBV (DNA ≥500 IU/mL) HCV (Ab+ with detectable RNA) HBV/HCV co-infection;
  5. History of neurologic/psychiatric disorders;
  6. Recent or current substance abuse;
  7. Prior allogeneic organ/hematopoietic stem cell transplantation.
* 4) Hypersensitivity to study drug or its excipients.
* 5) Active autoimmune disease requiring treatment or history within 2 years. Exceptions: Vitiligo/alopecia/psoriasis not needing systemic therapy Hypothyroidism managed only with hormone replacement Type 1 diabetes controlled solely with insulin.
* 6) Pregnant/lactating women;
* 7) Any uncontrolled systemic disease increasing study risk (per investigator);
* 8) Other unsuitable conditions determined by investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histologically or cytologically confirmed locally advanced or metastatic solid tumors with disease progression (radiographic or clinical) after ≥1 line of prior standard therapy, unsuitable for/intolerant to standard therapy.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Grade ≥3 irAEs | 2 years

SECONDARY OUTCOMES:
Incidence of adverse events | 2 years
Incidence of treatment-related adverse events | 2 years
Incidence of immune-related adverse events | 2 years

OTHER OUTCOMES:
Objective response rate | 2 years
Overall Survival | 2 years
Progression-Free Survival | 2 years
Disease Control Rate | 2 years
Duration of Response | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No